CLINICAL TRIAL: NCT06385860
Title: Research on the Prediction Model for Early Biliary Stasis After Bariatric Surgery Based on Machine Learning Algorithms
Brief Title: Prediction Model for Early Biliary Stasis After Bariatric Surgery
Acronym: PM-EBS-BS
Status: Not yet recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Wang Siqi, Principal Investigator, China-Japan Friendship Hospital
Other Study IDs: GTMGS0423
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Obesity; Diabetes; Gallstones; Biliary Stasis
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Gallstones; Cholestasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Developing and validating a predictive model to estimate the risk of early biliary stasis following bariatric surgery

DETAILED DESCRIPTION:
This study aims to create and validate a model that predicts the likelihood of early biliary stasis in obese patients following bariatric surgery (sleeve gastrectomy and Roux-en-Y gastric bypass)

ELIGIBILITY:
Inclusion Criteria:

1. BMI ≥32.5 kg/m2 with one or more obesity-related comorbidities.
2. BMI >35 kg/m2 without coexisting medical problems
3. complete preoperative and follow-up data.

Exclusion Criteria:

1. other bariatric procedures.
2. contraindications for bariatric surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to include patients who will undergo bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
early biliary stasis | one month
  The incidence of early biliary stasis after bariatric surgery
prediction model | six months
  Area under the curve (AUC) of the prediction model

IPD SHARING:
Plan to Share IPD: Undecided